CLINICAL TRIAL: NCT01557985
Title: Single Dose Pharmacokinetics and Pharmacodynamics of Bupivacaine Following Transversus Abdominis Plane (TAP) Block in Neonates
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: CMH IRB 2010-14308
Record Dates: First submitted 2012-03-13; First posted 2012-03-20 (Estimated); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain
Keywords: children; regional anesthesia; postoperative pain management; local anesthetic solution; toxicity
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transversus abdominis plane (TAP) Block: All participants in the study will receive a Transverses abdominis plane (TAP) Block in conjunction with their surgery.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — The volume of Bupivacaine per block will be 0.5 mL at 0.125%.

SUMMARY:
This study is being done to try to learn more about how a child's body breaks down bupivacaine, a local anesthetic medication that is being used for pain control. This study will provide information about how much medication gets into the bloodstream and how long it remains in the blood. Newborns and young infants often process drugs in their body in a different way than older children. This study will help the investigators determine how bupivacaine is broken down in the body of infants.

DETAILED DESCRIPTION:
A transverse abdominal plane (TAP_ block will be performed by one of the investigators who is adept in using ultrasound guidance after induction of general anesthesia. The dose of bupivacaine administered will be based on the weight of the patient. This dose is consistent with routine levels of local anesthetic used for peripheral nerve blocks and is lower than toxic levels so there will be no additional change in renal or liver function. Whole blood samples will be collected on a piece of filter paper from either an arterial, central, peripheral line or heel stick. The extracts from dried blood samples (DBS; calculated volume 20 µL) collected on filter paper will be analyzed using an LC-MS/MS system in combination with online extraction (LC/LC-MS/MS). Blood samples will be obtained at 0, 5, 15, 30, 60, 120 minutes, 4, 24, 48 hours. If obtained from a heel stick, these samples will be obtained at time of glucose sampling or a clinical indication. Subjects will be considered evaluable if they have 5 samples. All sampling for the study will be based on concurrent sampling so there will be no additional blood draws.

Pain will be assessed by the bedside nurse or study research assistant using the Neonatal Infant Pain Scale (NIPS). As part of the standard of care in this institution, nurses will have the opportunity to administer additional pain medications including but not limited to intravenous fentanyl or morphine. This will be done as per standing orders if the neonate meets criteria for additional analgesia, in other words, if there is an increase in pain as indicated by the NIPS pain scores. NIPS score will be recorded prior to each blood draw and every 8 hours while the subject is enrolled in the study. The NIPS will be the primary clinical outcome measure for this study. Blood pressure and heart rate will also be recorded as a physiologic correlate for drug level at these times.

ELIGIBILITY:
Inclusion Criteria:

* Neonates under 28 days of age undergoing any abdominal surgery including laparotomy, colostomy placement. In addition neonates who have procedures performed using laparoscopic as well as open techniques will be included
* Written informed consent from parent or guardian

Exclusion Criteria:

* Neonates with significant cardiovascular disease (any child with any congenital heart disease will be excluded from the study)
* Neonates with significant liver disease (any neonate with ALT/AST elevated 30% above normal values as determined by the lab at Lurie Children's at the time of testing)
* Neonates under 1.65 kg

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates younger than 28 days undergoing any abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Bupivacaine | Participants will be followed for the duration of anesthesia and after surgery, an average of 48 hours
  Cmax of bupivacaine in neonates undergoing the TAP block over a period of 48 hours

SECONDARY OUTCOMES:
Pharmacodynamics of Bupivacaine | participants will be followed for the duration of anesthesia and after surgery, an average of 48 hours
  Validated observational pain scale, Neonatal Infant Pain Scale (NIPS), as a clinical outcome correlate for bupivacaine levels

CONTACTS AND LOCATIONS:
Overall Officials: Santhanam Suresh, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Abdel-Rahman SM, Jacobs RF, Massarella J, Kauffman RE, Bradley JS, Kimko HC, Kearns GL, Shalayda K, Curtin C, Maldonado SD, Blumer JL. Single-dose pharmacokinetics of intravenous itraconazole and hydroxypropyl-beta-cyclodextrin in infants, children, and adolescents. Antimicrob Agents Chemother. 2007 Aug;51(8):2668-73. doi: 10.1128/AAC.00297-07. Epub 2007 May 21. PMID 17517842
- [Background] Bielsky A, Efrat R, Suresh S. Postoperative analgesia in neonates after major abdominal surgery: 'TAP' our way to success! Paediatr Anaesth. 2009 May;19(5):541-2. doi: 10.1111/j.1460-9592.2009.02988.x. No abstract available. PMID 19453587
- [Background] Zhang YL, Bendrick-Peart J, Strom T, Haschke M, Christians U. Development and validation of a high-throughput assay for quantification of the proliferation inhibitor ABT-578 using LC/LC-MS/MS in blood and tissue samples. Ther Drug Monit. 2005 Dec;27(6):770-8. doi: 10.1097/01.ftd.0000185766.52126.bd. PMID 16306853
- [Background] Frassetto L, Baluom M, Jacobsen W, Christians U, Roland ME, Stock PG, Carlson L, Benet LZ. Cyclosporine pharmacokinetics and dosing modifications in human immunodeficiency virus-infected liver and kidney transplant recipients. Transplantation. 2005 Jul 15;80(1):13-7. doi: 10.1097/01.tp.0000165111.09687.4e. PMID 16003227
- [Background] Christians U, Jacobsen W, Serkova N, Benet LZ, Vidal C, Sewing KF, Manns MP, Kirchner GI. Automated, fast and sensitive quantification of drugs in blood by liquid chromatography-mass spectrometry with on-line extraction: immunosuppressants. J Chromatogr B Biomed Sci Appl. 2000 Oct 1;748(1):41-53. doi: 10.1016/s0378-4347(00)00380-7. PMID 11092585
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140